CLINICAL TRIAL: NCT06726668
Title: Evaluation of the Role of Ultrasonographic Subclavian Vein Collapsibility Index in Estimating Fluid Requirement in Shocked Traumatic Patients in Emergency Department at Assiut University Hospital
Brief Title: Estimating Fluid Requirement in Shocked Traumatic Patients by US on SCV
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Abdelhameed, Emergency medicine resident physician at Assiut University Hospitals, Assiut University
Other Study IDs: US Subclavian vein Shock
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Shock; Trauma
Keywords: Us; Subclavian vein; Shock; Trauma
MeSH Terms: conditions — Shock; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research question Is the ultrasonographic SCV collapsability index effective in estimating fluid requirements in shocked traumatic Patients ?

Purpose of the study To evaluate the effectiveness of ultrasonograghic SCV collapsibility index before and after the first hour of resuscitation in estimating the First 24 h of fluid requirement in shocked traumatic patients.

DETAILED DESCRIPTION:
Hypovolemic shock is a circulatory malfunction associated with inadequate tissue perfusion that leads to multi organ failure. Since it results from either blood Loss or extracellular fluid loss, quick onset hypovolemia is usually the cause. Blood loss-related hypovolemic shock is known as hemorrhagic shock. Hemorrhagic shock is typically the primary cause of shock in trauma victims, while numerous other conditions can also contribute to shock. Hemorrhage accounts for 30 to 40% of trauma-related deaths, of which 33 to 56% happen in the prehospital phase and over 40% happen in the first 24 h. This means that it can be lethal very quickly. Hematocrit levels, biochemical markers, physical examination results, and other conventional measures are used to identify hypovolemia, but are not precise markers or trustworthy since they can be deemed normal when the body's compensatory mechanisms kick in, which could cause delays in the identification of volume loss. While tachycardia is a symptom of acute fluid loss, its sensitivity and specificity are insufficient for diagnosis or monitoring because it can be altered by a variety of internal and external signals. As A central line is an invasive procedure with potential complications (venous thrombosis, infection, pneumothorax, arterial puncture) during or after the procedure and poor predictive value, measurement of CVP is not practically used in hypovolemic patients admitted to the emergency department (ED). Focused assessment with sonography for trauma (FAST) has shown to be an effective way to identify bleeding sites in trauma patients using sonography. FAST took an average of 4 min per patient and was used successfully as a primary screening procedure at the hospital's entrance for traumatized mass casual patients. However, it provides no information regarding the patient's hemodynamic status, blood loss, amount lost, or response to resuscitation. As such, we require techniques for early detection of hypovolemia and accurate follow-up. The use of ultrasonography in critical care has grown in recent years due to technological advancements. The SCV is widely acknowledged as a trustworthy metric for assessing hemodynamic conditions. When the body experiences volume loss, the compensatory vasoconstrictor reaction has little effect on the SCV diameter. The noninvasive quick diagnosis, and low cost of sonographic measurement Of SCV diameter make this method a valuable tool for determining fluid requirements and evaluating Volume status in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic patients who will come to emergency department at Assiut university Hospital between march 2025 to march 2026 and will be admitted after stabilization to the Inpatient ward or ICU

Exclusion Criteria:

* Patients or their Relatives refuse participation in the study.

  * Patients who will be transferred to another hospital

    * • Pregnant women.
  * Age below 18 and more than 60.
  * Failure of follow-up of any patient.
  * Cardiopulmonary resuscitation on arrival.
  * Contraindicating fluid challenges, such as cardiac insufficiency and Renal failure .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Total coverage sample of all traumatic patients who will be admitted to emergency department Assiut university who fulfill the inclusion criteria during study period of 12 months from 1st of March 2025 to 1st of March 2026.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To estimate and predict the fluid requirement using ultrasonograghic Sub Clavian vein collapsibility index before and after the first hour of resuscitation | Before resuscitation and after 1 hour of resuscitation
  In the first hour of resuscitation, the patients (unstable shocked) will be given 1 L of crystalloid solution for fluid resuscitation ( according to recent ATLS guidelines). If the patient is still unstable after 1 Liter of fluid or had ongoing blood loss, O- negative blood transfusion will be administered and type-specific blood Will be ordered and the trauma team activated massive transfusion protocol according to recent ATLS Guidelines even if normal hemoglobin.
  The traumatic patients after 1 h of resuscitation were divided into two groups (SCV non -Repleted) and (SCV Repleted) group as (if thereis still an SCV diameter of < 7 mm after the first hour of resuscitation they are called (the SCV non -Repleted) group. And if the SCV diameter of ≥ 7 mm after the first hour of resuscitation) they are called the (SCV Repleted) group.

SECONDARY OUTCOMES:
To estimate and predict the First 24-h fluid requirement using repeated ultrasonograghic SCV collapsibility index. | In the first 24 hours of resuscitation
  In this study, it's predicted that after the first hour of resuscitation (the SCV non - Repleted) group needed more than 1-2 ml/kg/hour in the first24 hours (more than 2400 ml fluid), and the (SCV Repleted) group we predict that after the first hour of resuscitation, they will need the average 1-2 ml/kg/hr. (average 2400 ml fluid) or less in the first 24 h. Patients will be clinically assessed and managed as per the ABC protocol.
-To assess the role of ultrasonograghic SCV CI in rapidly detecting early shock stages. | In the first 24 hours of resuscitation
  Traumatic patients will be considered shocked if they have signs of shock such as decreased blood pressure < 90/60 mmHg , heart rate > 100 b/m, cold clammy skin, capillary refill > 2 s and their shock index above0.9.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Mohamed Abdelhameed, Resident, Principal Investigator
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided